CLINICAL TRIAL: NCT01521650
Title: Probiotics for Reduction of Colonisation With Pathogenic Bacteria in the Oropharynx in Connection With Anaesthesia
Brief Title: Probiotics Against Pathogenic Bacteria in Connection With Anaesthesia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Region Skane (Other)
Collaborators: Lund University (Other)
Responsible Party: Principal Investigator, Bengt Klarin, MD Consultant, Region Skane
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: ProAnest
Record Dates: First submitted 2012-01-26; First posted 2012-01-31 (Estimated); Last update posted 2021-03-10 (Actual); Status verified 2021-03

CONDITIONS: Oropharyngeal Microbiology
Keywords: Probiotics; Anaesthesia; Intubation; Pathogenic bacteria
MeSH Terms: interventions — Probiotics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Probiotics (Experimental): Patients will gurgle and swallow a mixture of probiotic bacteria
  Interventions: Dietary Supplement: Probiotics
- Control (No Intervention): No intervention. What has been the standard procedure so far

INTERVENTIONS:
Dietary Supplement: Probiotics — Patients will gurgle and swallow a mixture of probiotic bacteria
  Other Names: Lactobacillus plantarum 299; Lactobacillus plantarum 299v
  Arms: Probiotics

SUMMARY:
Longer surgical procedures require intubation and there is a potential risk of contaminating the lower airways with pathogenic bacteria from the mouth and oropharynx.

Healthy people seldom have pathogenic bacteria originating from the gastro-intestinal canal but those do occur among patients, both in those not so sick and patients with more severe problems.

For ICU patients we have seen a reduction of emerging enteric bacteria in patients given oral care with probiotics and this is a pilot study to explore the possibility of the same kind of positive effects in patients due for longer (more than 4 hours of anesthesia) procedures.

Randomisation

* No prophylaxis
* Preparation with a probiotic suspension before intubation.

Cultures

* oropharynx

  * before treatment
  * after intubation
  * before extubation
  * day 1 postoperatively
* tracheal secretions

  * after intubation
  * before extubation

ELIGIBILITY:
Inclusion Criteria:

* Adult patients
* Planned interventions
* Anaesthesia > 4 hours and requiring intubation

Exclusion Criteria:

* Ulcers in the mouth, oropharynx, oesophagus and stomach
* Current infections in the airways
* Known immuno deficiences
* Emergency cases

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2012-01; Primary Completion 2019-03 (Actual); Study Completion 2020-07 (Actual)

PRIMARY OUTCOMES:
Differences in pathogenic bacteria in the oropharynx and lower airways | During hospitalization, up to 4 weeks
  Emerging and resident bacteria will be compared for the cultures taken in the oropharynx and from tracheal secretions in conection with anaestesia and a surgical intervention

SECONDARY OUTCOMES:
White blood cells | During hospitalization, up to 4 weeks
  WBC taken pre-op and days 1,2,3 post-op
CRP | During hospitalization, up to 4 weeks
  CRP taken pre-op and days 1,2,3 post-op
Pneumonia | Up till 7 days postoperatively
  X-ray verified infiltrations in combination with expectorates
Length of hospital stay | time to discharged from hospital or patients death
  Comparison of length of stay between the intervention group and the control group

CONTACTS AND LOCATIONS:
Overall Officials: Bengt klarin, MD PhD, Principal Investigator — Lund University
Locations (1):
- Lund University Hospital, Lund, Sweden

IPD SHARING:
Plan to Share IPD: Yes
Results are intended to be published in a scientific journal

REFERENCES:
- [Background] Stjernquist-Desatnik A, Warfving H, Johansson ML. Persistence of Lactobacillus plantarum DSM 9843 on human tonsillar surface after oral administration in fermented oatmeal gruel. A pilot study. Acta Otolaryngol Suppl. 2000;543:215-9. doi: 10.1080/000164800454422. PMID 10909023
- [Background] Klarin B, Molin G, Jeppsson B, Larsson A. Use of the probiotic Lactobacillus plantarum 299 to reduce pathogenic bacteria in the oropharynx of intubated patients: a randomised controlled open pilot study. Crit Care. 2008;12(6):R136. doi: 10.1186/cc7109. Epub 2008 Nov 6. PMID 18990201